CLINICAL TRIAL: NCT04530409
Title: Timing of Corticosteroids in COVID-19, II. Post COVID-19 Follow-up
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ClinAmygate (Other)
Responsible Party: Principal Investigator, Emad R Issak, Dr, ClinAmygate
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR0012
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Covid19; Corticosteroids
Keywords: COVID19; dexamethazone; methylpredisolone; early recovery
MeSH Terms: conditions — COVID-19 | interventions — Dexamethasone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early CS (Experimental): early use of dexamethasone as early as the laboratory confirmation of inflammation.
  Interventions: Drug: Early-Corticosteroids
- Late CS (No Intervention): Dexamethasone is to be used lately upon the deterioration of cases i.e. sPO2 < 92%

INTERVENTIONS:
Drug: Early-Corticosteroids — early use of dexamethasone/Methylprednisolone as early as laboratory evidence of high inflammatory markers
  Other Names: Dexamethasone; Methylprednisolone
  Arms: Early CS

SUMMARY:
Timing of of corticosteroids administration is very important in COVID19 cases for the recovery and decrease the mortality.

DETAILED DESCRIPTION:
The sickest patients with COVID-19 suffer a hyperinflammatory state-a cytokine storm-that has features in common with a rare haematological condition called haemophagocytic lymphohistiocytosis. Immune suppression should help such patients. By contrast, immune suppression during the early phase of the viral infection might allow increased viral replication and aggravate the disease.

The 3C-like proteinase on SARS-CoV-2 (nsp5) inhibits HDAC2 transport into the nucleus, and so impairs the way in which it mediates inflammation and cytokine responses, so activation of histone deacetylase by dexamethasone may directly oppose the action of SARS-CoV-2.

Timing of of corticosteroids administration is very important in COVID19 cases for the recovery and decrease the mortality.

ELIGIBILITY:
Inclusion Criteria:

* any case with COVID-19 more than or equal to 18 years
* mild and moderate severity

Exclusion Criteria:

* Severe to critical COVID-19
* Any contra-indication for the interventional drug
* Mentally disabled cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of cases that will need hospitalization | 10 days
  Deterioration in the clinical picture of cases that necessitate hospitalization
Percentage of cases that will need oxygen supplementation | 10 days
  Percentage of cases whose clinical status deteriorate that their sPO2 become less than 92%
28-days mortality | 28 days
  Percentage of cases who died within 28 days of presentation

SECONDARY OUTCOMES:
Percentages of COVID-19 Severity according to CDC 2020 | 10 days
  Percentages of COVID-19 severity according to CDC 2020
Time to return to daily activity | 60 days
  Time to return to daily activity level
Percentage of cases with increased d-dimer | 10 days
  Percentage of cases with increased d-dimer from baseline
Percentage reduction in CRP | 10 days
  Percentage reduction in CRP from baseline
Percentage reduction in LDH | 10 days
  Percentage reduction in LDH from baseline
Percentage reduction in Ferritin | 10 days
  Percentage reduction in Ferritin from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Emad R Issak, Principal Investigator — Assalam Clinics
Locations (1):
- Asalam, Maadi, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spoorenberg SM, Deneer VH, Grutters JC, Pulles AE, Voorn GP, Rijkers GT, Bos WJ, van de Garde EM. Pharmacokinetics of oral vs. intravenous dexamethasone in patients hospitalized with community-acquired pneumonia. Br J Clin Pharmacol. 2014 Jul;78(1):78-83. doi: 10.1111/bcp.12295. PMID 24400953